CLINICAL TRIAL: NCT03447548
Title: Neurofeedback Processing Speed Training to Improve Social Functioning in Teenagers and Young Adults at Clinical High Risk for Psychosis
Brief Title: Neurofeedback Training for High Risk Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HHC-2017-0190; 1R33MH111850-01A1 (NIH)
Record Dates: First submitted 2018-01-15; First posted 2018-02-27 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Prodromal Schizophrenia
Keywords: Cognitive training; Social function; Processing speed
MeSH Terms: conditions — Schizotypal Personality Disorder; Social Adjustment

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with intervention versus active control
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Processing speed training (Experimental): Neurofeedback processing speed training
  Interventions: Behavioral: Neurofeedback processing speed training
- Active control (Active Comparator): Computer games
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: Neurofeedback processing speed training — Processing speed training on tablets that incorporates changes in pupil size to titrate the learning algorithm
  Arms: Processing speed training
Behavioral: Active control — Commercially available games on tablet
  Arms: Active control

SUMMARY:
Young people who are at great risk for developing psychosis have cognitive deficits which are strongly related to functioning in the community. This study looks to target a specific cognitive skill called processing speed to see if improving the ability to process information in a timely manner will improve social function in adolescents and young adults at risk for developing schizophrenia. Half will receive neurofeedback cognitive training targeting processing speed while the other half will receive an active control.

DETAILED DESCRIPTION:
Processing speed deficits are characteristic of schizophrenia and related to its functional impairment, including in its nascent stages, during a putatively prodromal or clinical high risk period. These cognitive deficits have proven relatively refractory to pharmacologic strategies, though the deficits can be improved with cognitive remediation programs in schizophrenia. The cognitive gains can then generalize to functional improvement, particularly early in the course of illness (i.e. first episode psychosis). Although processing speed deficits are also prevalent in young people identified as at clinical high risk for psychosis (i.e. "psychosis risk syndrome"), and related to their concurrent impaired function and predictive of later psychosis (onset of which occurs in 20-25% of clinical high risk cohorts), little research has focused on how to remediate these deficits in clinical high risk patients. Remediating core cognitive deficits in clinical high risk patients could plausibly address present functional impairment in these young people and moderate illness progression. The investigators propose to conduct a double-blind randomized trial in 105 clinical high risk patients to examine a focal processing speed training program versus an active control in terms of improvement in processing speed and social function, and reduction in prodromal symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Case identification and ascertainment depends on the fulfillment of the Criteria of Prodromal States as evaluated using the Structured Interview for Prodromal Syndromes: (1) attenuated positive symptom state which includes the emergence or worsening over the past year of non-psychotic disturbances in thought content, thought process or perceptual abnormality, (2) brief intermittent positive symptoms, and (3) genetic risk and deterioration.
* Processing speed at least 0.5 Standard Deviation below the norm, as indexed by baseline performance on Digit Symbol Coding of 8 or below
* Age range 12-25 (this age range also comprises the main period of risk for psychosis)
* Written informed consent by patients >18 years old, and written assent by subjects <18 years old, with written informed consent by both parents (unless one is deceased or unavailable). Participants who turn 18 while in the study will be re-consented as adults through written informed consent.

Exclusion Criteria:

* Current or past diagnosis of psychotic disorder noted at baseline assessment (schizophrenia, schizophreniform, bipolar, schizoaffective, major depression with psychotic features, substance-induced psychosis, psychosis due to a medical condition.
* Neurological, neuroendocrine or major medical disorders: as putative prodromal symptoms could be secondary to these and unrelated to risk for primary psychotic disorders (clinical interview), including seizure disorder and history of significant traumatic brain injury
* Intelligence Quotient < 70: as putative prodromal symptoms could be secondary to these and unrelated to risk for primary psychotic disorders
* Positive symptoms that occur only in the context of substance abuse or withdrawal (i.e. within one month), so as not to include those at risk for substance-induced psychotic disorder
* Lack of fluency in English: subjects must speak English to complete behavioral assessments for which psychometric properties have been established in English, complete cognitive training, and in order to comprehend and comply with protocol requirements.
* Substance abuse or dependence (including alcohol and marijuana) in previous six months: for purposes of standardization and interpretation of cognitive data.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change on the Wechsler Intelligence Scale Processing Speed Index | Baseline, 1 month, 2 month, 6 month
  Change on a paper and pencil test of processing speed

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Connecting Adolescents with Psychosis (CAP), Child & Adolescents Day Program, Hartford, Connecticut
  - Olin Neuropsychiatry Research Center, Hartford, Connecticut